CLINICAL TRIAL: NCT05622045
Title: Does Personality Predict Patient Adherence, Health Behaviors, and Weight Loss Outcomes During the Latino Crossover Semaglutide Study (LCSS)? (Story-LCSS Project)
Acronym: StoryLCSS
Status: Active, not recruiting | Type: Observational
Sponsor: Loma Linda University (Other)
Collaborators: Scaled Insights (Industry)
Responsible Party: Sponsor
Other Study IDs: 5220330
Record Dates: First submitted 2022-11-07; First posted 2022-11-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Body Weight Changes
Keywords: artificial intelligence; obesity; weight loss
MeSH Terms: conditions — Obesity; Body Weight Changes; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Story-LCSS
  Interventions: Behavioral: Voice data

INTERVENTIONS:
Behavioral: Voice data — Recorded response to a question about their participation in a weight loss study.

SUMMARY:
The goal of this observational study is to learn about the personality attributes and values of people living with obesity that are part of the Latino community, and how these personality attributes and values can help to predict success during a weight loss program.

The main questions it aims to answer are:

* What are the personality attributes and values of people living with obesity that sign up to the LCSS-Latino Crossover Semaglutide Study trial?
* Can behavioral artificial intelligence (a computer formula) predict which patients will complete the LCSS-Latino Crossover Semaglutide Study trial?
* How do behavioral artificial Intelligence predictions (a computer formula) compare to clinician predictions of patient success?
* Can behavioral artificial intelligence (a computer formula) predict patient weight loss, calorie consumption and physical activity levels during the LCSS-Latino Crossover Semaglutide Study trial? Participants will be recorded in English and Spanish while responding to a question regarding participation in a weight loss study.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the LCSS-Latino Crossover Semaglutide Study

Exclusion Criteria:

* Not a participant of the LCSS-Latino Crossover Semaglutide Study at the point of data collection

Ages: 18 Years to 74 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hispanic men and women, 18 to 74 years of age, with obesity, residing in Southern California, who are taking part in the LCSS-Latino Crossover Semaglutide Study.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Predicted patient weight change success | The voice data measurement will take place at baseline and take about 10-15 minutes for collection to take place.
  Predicted patient weight change as determined by Scaled Insights Behavioural Artificial Intelligence based on subject voice data. Weight loss exceeding 5-10 pounds over 6 months will be considered to be successful. Predicted weight change will be compared to the weight change measured in a separate clinical trial [Latino Crossover Semaglutide Study (LCSS) NCT05087342]. Similar weight change values between the predicted and measured outcomes will indicate that the Scaled Insights Behavioural Artificial Intelligence is good predictor.
Clinician predictions | The clinician judgement will be measured during the second month of the subject's weight loss study.
  Clinician (physician) judgement of patient weight loss success during a weight loss study.
Predicated patient calorie intake | The voice data measurement will take place during the subject's initial clinic visit and take about 10-15 minutes for collection to take place.
  Predicted patient calorie intake as determined by Scaled Insights Behavioural Artificial Intelligence based on subject voice data. Predicted calorie intake will be compared to the calorie intake measured in a separate clinical trial [Latino Crossover Semaglutide Study (LCSS) NCT05087342]. Similar calorie values between the predicted and measured outcomes will indicate that the Scaled Insights Behavioural Artificial Intelligence is good predictor.
Predicated patient physical activity level | The voice data measurement will take at baseline and take about 10-15 minutes for collection to take place.
  Predicted patient physical activity level as determined by Scaled Insights Behavioural Artificial Intelligence based on subject voice data. Predicted physical activity will be compared to the physical activity measured in a separate clinical trial [Latino Crossover Semaglutide Study (LCSS) NCT05087342]. Similar physical activity level values between the predicted and measured outcomes will indicate that the Scaled Insights Behavioural Artificial Intelligence is good predictor.

SECONDARY OUTCOMES:
Personality attributes and values | The voice data measurement will take place at baseline and take about 10-15 minutes for collection to take place.
  Extrapolated personality attributes and values as determined by Scaled Insights Behavioural Artificial Intelligence based on subject voice data. These are qualitative non-numerical descriptors.
Predicted patient attrition rate | The voice data measurement will take place at baseline and take about 10-15 minutes for collection to take place.
  Predicted patient attrition rate from the weight loss study as determined by Scaled Insights Behavioural Artificial Intelligence based on subject voice data. Predicted patient attrition rate will be compared to the attrition rate occurring during the weight loss study. Similar attrition rates between the predicted and actual rates will indicate that the Scaled Insights Behavioural Artificial Intelligence is good predictor.

CONTACTS AND LOCATIONS:
Overall Officials: Celine Heskey, DrPH, Principal Investigator — Loma Linda University
Locations (1):
- Nutrition Research Center, School of Public Health, Loma Linda University, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
There is not plan currently to share IPD outside of the collaborators that are part of the study. It is possible that requests may be made by students later on to use data for secondary data analysis as part of their academic research projects, and the research collaborators will decide if unidentified IPD would be shared at such a time.

REFERENCES:
- [Background] Alberga AS, Russell-Mayhew S, von Ranson KM, McLaren L. Weight bias: a call to action. J Eat Disord. 2016 Nov 7;4:34. doi: 10.1186/s40337-016-0112-4. eCollection 2016. PMID 27826445
- [Background] Dalle Grave R, Calugi S, Compare A, El Ghoch M, Petroni ML, Tomasi F, Mazzali G, Marchesini G. Weight Loss Expectations and Attrition in Treatment-Seeking Obese Women. Obes Facts. 2015;8(5):311-8. doi: 10.1159/000441366. Epub 2015 Oct 8. PMID 26444382
- [Background] Flint SW, Leaver M, Griffiths A, Kaykanloo M. Disparate healthcare experiences of people living with overweight or obesity in England. EClinicalMedicine. 2021 Sep 15;41:101140. doi: 10.1016/j.eclinm.2021.101140. eCollection 2021 Nov. PMID 34585130
- [Background] Flint SW, Piotrkowicz A, Watts K. Use of Artificial Intelligence to understand adults' thoughts and behaviours relating to COVID-19. Perspect Public Health. 2022 May;142(3):167-174. doi: 10.1177/1757913920979332. Epub 2021 Jan 21. PMID 33472547
- [Background] Hardcastle SJ, Taylor AH, Bailey MP, Harley RA, Hagger MS. Effectiveness of a motivational interviewing intervention on weight loss, physical activity and cardiovascular disease risk factors: a randomised controlled trial with a 12-month post-intervention follow-up. Int J Behav Nutr Phys Act. 2013 Mar 28;10:40. doi: 10.1186/1479-5868-10-40. PMID 23537492
- [Background] Puhl RM, Phelan SM, Nadglowski J, Kyle TK. Overcoming Weight Bias in the Management of Patients With Diabetes and Obesity. Clin Diabetes. 2016 Jan;34(1):44-50. doi: 10.2337/diaclin.34.1.44. No abstract available. PMID 26807008
- [Background] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185